CLINICAL TRIAL: NCT04020055
Title: An Open-label Study to Evaluate the Safety and Pharmacokinetics of Migalastat HCl in Subjects With Fabry Disease and Amenable GLA Variants and Severe Renal Impairment or End-Stage Renal Disease Treated With Hemodialysis
Brief Title: A Study to Evaluate Migalastat in Fabry Subjects With Amenable GLA Variant and Renal Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT1001-025
Expanded Access: NCT01476163 (Available)
Record Dates: First submitted 2019-06-24; First posted 2019-07-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Fabry Disease
Keywords: Renal Disease; Severe Renal Impairment (SRI); End-Stage Renal Disease (ESRD)
MeSH Terms: conditions — Fabry Disease; Kidney Diseases; Renal Insufficiency; Kidney Failure, Chronic | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Severe Renal Impairment (Experimental): All subjects will receive migalastat 123 mg, equivalent to 150 mg migalastat HCl (hereafter, migalastat) at a dose regimen based on their eGFRMDRD result at Visit 1. Subjects will take 1 migalastat capsule orally with water either every 4 or 7 days.
- Cohort 2: End-Stage Renal Disease (Experimental): All hemodialysis subjects will receive migalastat 123 mg, equivalent to 150 mg migalastat HCl (hereafter, migalastat). Subjects will take 1 migalastat capsule orally with water every other week.
  Interventions: Drug: migalastat HCl 150 mg

INTERVENTIONS:
Drug: migalastat HCl 150 mg — migalastat HCl 150 mg capsule
  Other Names: migalastat; AT1001
  Arms: Cohort 2: End-Stage Renal Disease

SUMMARY:
An Open-label Study to Evaluate the Safety and Pharmacokinetics of Migalastat HCl in Subjects with Fabry Disease and Amenable GLA Variants and Severe Renal Impairment (SRI) or End Stage Renal Disease (ESRD)

DETAILED DESCRIPTION:
This is an open-label, non-comparative study for subjects with Fabry disease who have an estimated glomerular filtration rate (eGFR) based on the Modification of Diet in Renal Disease equation (eGFRMDRD) value of < 30 mL/min/1.73 m2. Subjects may have had previous exposure to migalastat, either commercially or as a participant in a previous migalastat study.

Two distinct populations of subjects with Fabry disease and renal impairment will be enrolled into this study:

* Cohort 1: Subjects with SRI not receiving any type of dialysis treatment
* Cohort 2: ESRD subjects who are receiving hemodialysis treatment, either standard hemodialysis (HD) or hemodiafiltration (HDF). Only subjects who can receive HD/HDF at the study clinic or at an affiliated center where the Investigator already has oversight should be enrolled into Cohort 2.

Subjects entering into this study will undergo screening (Visit 1) to confirm enrollment eligibility including confirmatory GLA genotyping. Subjects who meet eligibility criteria will have a Baseline Visit (Visit 2) within 30 days of screening. Subjects who do not meet eligibility criteria (eg, subjects with an eGFR > 30 mL/min/1.73 m2) may be re-screened.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older, diagnosed with Fabry disease.
2. Subject (or legally authorized representative as applicable) is willing and able to provide written informed consent and authorization for use and disclosure of Personal Health Information
3. Subject has a GLA variant that is amenable to migalastat recorded in their medical records
4. Subject has at least 1 documented eGFR value of < 30 mL/min/1.73 m2 within the last 3 months and has an eGFRMDRD value of < 30 mL/min/1.73 m2 at Visit 1
5. Subjects with ESRD have been on a stable 2- or 3-times a week HD (standard or HDF) regimen for at least 2 months prior to the screening visit
6. Subjects with ESRD must commit to completing at least 4 standard HD or HDF sessions during each 2-week dosing interval.
7. Subjects with ESRD must commit to completing the entire prescribed duration for each dialysis session.
8. If of reproductive potential, both male and female patients agree to use a medically accepted method of contraception

Exclusion Criteria:

1. Subject has undergone kidney transplantation
2. Subject is on peritoneal dialysis
3. Subject is treated or has been treated with another investigational drug (except migalastat) within the 30 days
4. Subject has undergone any gene therapy at any time prior to the study or anticipates undergoing gene therapy during the study.
5. Subject has had a documented transient ischemic attack, stroke, unstable angina, or myocardial infarction
6. Subject has clinically significant unstable cardiac disease
7. Subject has any intercurrent illness or condition that may preclude the subject from fulfilling the protocol requirements
8. Subject has a history of allergy or sensitivity to migalastat (including excipients) or other iminosugars (eg, miglustat, miglitol)
9. Subject requires concurrent treatment with Glyset® (miglitol), Replagal® (agalsidase alfa), or Fabrazyme® (agalsidase beta)
10. Subject requires concurrent treatment with Zavesca® (miglustat) or has been treated with Zavesca
11. Female subject is pregnant or breast-feeding
12. Subject is unable to comply with study requirements
13. In France only, protected persons as defined by the Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Time to maximum concentration (tmax) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Apparent terminal elimination half-life (t½) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK
Concentration at the end of a dosing interval at steady state (Ctrough) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Average plasma migalastat concentration over the dosing interval (Cavg) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Area under the concentration-time curve at steady state during the dosing interval (AUC0-τ) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Area under the concentration-time curve from zero time (pre-dose) extrapolated to infinite time (AUC0-∞) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Apparent plasma clearance (CL/F) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK
Apparent terminal phase volume of distribution (Vz/F) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Dialysis clearance (CLD) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Volume of dialysate collected during the interval (VD) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Mean migalastat concentration in dialysate (CD) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Amount recovered in dialysate (AeD) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Fraction of the dose recovered in dialysate (FeD) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Mean migalastat plasma concentration during the dialysis interval (P) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Mean inlet area under the curve (AUCinlet) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Mean outlet area under the curve (AUCoutlet) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Extraction ratio (ED) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Dialyzer blood flow (QD) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Cumulative amount excreted over all collection intervals (Ae0-τ) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Fraction of the dose recovered after the last measurable time point postdose (Fe0-τ) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.
Renal clearance (CLr) | Baseline through Month 12
  To characterize the pharmacokinetics (PK) of migalastat and validate the population PK (popPK) model and simulations.

SECONDARY OUTCOMES:
Adverse events (AEs) | Baseline through Month 12
  To assess the safety and tolerability of migalastat in Fabry subjects with severe renal impairment and end stage renal disease.
Change from baseline in estimated glomerular filtration rate (eGFR) based on the Modification of Diet in Renal Disease equation (eGFR MDRD) | Baseline through Month 12
  To assess the safety and tolerability of migalastat in Fabry subjects with severe renal impairment and end stage renal disease
Change from baseline eGFR based on the Chronic Kidney Disease Epidemiology Collaboration equation (eGFRCKD-EPI) | Baseline through Month 12
  To assess the safety and tolerability of migalastat in Fabry subjects with severe renal impairment and end stage renal disease
Change from baseline in plasma globotriaosylsphingosine (lyso-Gb3) | Baseline through Month 12
  To evaluate the pharmacodynamics (PD) of migalastat in subjects with Fabry disease and severe renal impairment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research, Study Director — Amicus Therapeutics
Locations (12):
- United States (3):
  - Emory University, Atlanta, Georgia
  - The Cleveland Clinic, Cleveland, Ohio
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc, Fairfax, Virginia
- Australia (2):
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Washington
- Japan (2):
  - Osaka University Hospital, Suita, Osaka
  - Shizuoka General Hospital, Shizuoka, Shizuoka
- Centro Hospitalar e Universitário de Coimbra (CHUC), Coimbra, Portugal
- Spain (3):
  - Hospital Universitari(o) de Bellvitge (HUB) Feixa Llarga, Barcelona
  - Hospital General Universitario de Elda, Elda
  - Hospital General Universitario Gregorio Marañon, Madrid
- Salford Royal Hospital, Salford, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No